CLINICAL TRIAL: NCT04361110
Title: Preoperative Findings on Non-specific CT in Patients With Primary Acute Intestinal Ischaemia; a Case-control Study
Brief Title: Radiological Findings in Primary Intestinal Ischaemia
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, David Straarup, Principal Investigator, Aalborg University Hospital
Other Study IDs: Acute intestinal ischaemia
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Acute Intestinal Ischemia
Keywords: Diagnoses Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Acute intestinal ischaemia: Abdominal CT scan within 48 hours preoperative.
  Interventions: Radiation: Computerized tomography scan of the abdomen
- Controls: Abdominal CT scan within 48 hours preoperative.
  Interventions: Radiation: Computerized tomography scan of the abdomen

INTERVENTIONS:
Radiation: Computerized tomography scan of the abdomen — Non-specific abdominal ct´s with different phases and contrast +/-.

SUMMARY:
To investigate which findings on a non-specific CT scan that predict acute primary intestinal ischaemia.

DETAILED DESCRIPTION:
48 patients with primary intestinal ischemia admitted in 4 consecutive years (2006-2009) in Department of Gastrointestinal Surgery, Aalborg University Hospital. Control group consists of 82 patients operated in the same department and in the same time range.

Abdominal CT scans are described with respect to intestinal diameter, changes in intestinal wall, extra intestinal changes and vessel pathology.

ELIGIBILITY:
Inclusion Criteria:

* Primary acute intestinal ischaemia in an abdominal operation.
* CT-scan within 48 hours preoperative.

Exclusion Criteria:

* Secondary intestinal ischaemia
* Intestinal ischaemia isolated intestinal mucosa.
* No CT-scan within 48 hours preoperative

Max Age: 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All operated patients at Department of Gastrointestinal surgery, Aalborg University Hospital, Denmark.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2009-12-31 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Intestinal wall pathology | 48 hours
  Incidense of CT findings in the radiological main group called "Intestinal wall pathology"
Gastrointestinal vessel pathology | 48 hours
  Incidense of CT findings in the radiological main group called "Gastrointestinal vessel pathologypathology"
Intestinal diameter | 48 hours
  Incidense of CT findings in the radiological main group called "Intestinal diameter"
Extraintestinal pathology | 48 hours
  Incidense of CT findings in the radiological main group called "Extraintestinal pathology"

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Menke J. Diagnostic accuracy of multidetector CT in acute mesenteric ischemia: systematic review and meta-analysis. Radiology. 2010 Jul;256(1):93-101. doi: 10.1148/radiol.10091938. PMID 20574087
- [Background] Karkkainen JM, Acosta S. Acute mesenteric ischemia (part I) - Incidence, etiologies, and how to improve early diagnosis. Best Pract Res Clin Gastroenterol. 2017 Feb;31(1):15-25. doi: 10.1016/j.bpg.2016.10.018. Epub 2017 Jan 4. PMID 28395784
- [Background] Tilsed JV, Casamassima A, Kurihara H, Mariani D, Martinez I, Pereira J, Ponchietti L, Shamiyeh A, Al-Ayoubi F, Barco LA, Ceolin M, D'Almeida AJ, Hilario S, Olavarria AL, Ozmen MM, Pinheiro LF, Poeze M, Triantos G, Fuentes FT, Sierra SU, Soreide K, Yanar H. ESTES guidelines: acute mesenteric ischaemia. Eur J Trauma Emerg Surg. 2016 Apr;42(2):253-70. doi: 10.1007/s00068-016-0634-0. PMID 26820988
- [Background] Cudnik MT, Darbha S, Jones J, Macedo J, Stockton SW, Hiestand BC. The diagnosis of acute mesenteric ischemia: A systematic review and meta-analysis. Acad Emerg Med. 2013 Nov;20(11):1087-100. doi: 10.1111/acem.12254. PMID 24238311
- [Background] Aschoff AJ, Stuber G, Becker BW, Hoffmann MH, Schmitz BL, Schelzig H, Jaeckle T. Evaluation of acute mesenteric ischemia: accuracy of biphasic mesenteric multi-detector CT angiography. Abdom Imaging. 2009 May-Jun;34(3):345-57. doi: 10.1007/s00261-008-9392-8. PMID 18425546
- [Derived] Straarup D, Gotschalck KA, Mikalone R, Thorlacius-Ussing O. Preoperative findings on non-specific CT in patients with primary acute intestinal ischemia: a case-control study. Eur J Trauma Emerg Surg. 2022 Aug;48(4):3025-3032. doi: 10.1007/s00068-021-01741-w. Epub 2021 Jul 3. PMID 34216221